CLINICAL TRIAL: NCT00401297
Title: Intervenable Host- Leishmania (Vianna) Interactions Project 3: Immune and Inflammatory Responses in L. (Viannia) Infection Aim 1: To Determine if Th1/Th2 Polarization Occurs and is Linked to the Outcome of Infection by L. Viannia
Brief Title: Th1/Th2 Polarization and Linkage to L. Viannia Infection Outcomes
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Dr. Diane McMahon-Pratt, Yale University
Other Study IDs: 0608001741; U19AI065866 (NIH)
Record Dates: First submitted 2006-11-16; First posted 2006-11-20 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2011-08

CONDITIONS: Leishmaniasis
Keywords: Leishmaniasis; L. Viannia; Leishmania; Colombia
MeSH Terms: conditions — Leishmaniasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine what types of cells participate in the defense of humans against Leishmania (skin parasites). People 18-70 years of age who have leishmaniasis, have healed leishmanial lesions, or are healthy are being invited to participate in this study. Approximately 150 people will participate in the study. Participants will be asked to provide some general information about themselves and about skin sores, if they have any. A skin test will be performed and a blood sample will be obtained. This study involves up to 3 visits; the first visit will last up to 5 hours and the second visit will last for 30 minutes. The third visit may be scheduled within 3 days after the second visit.

DETAILED DESCRIPTION:
The purpose of this study is to determine if Th1/Th2 polarization occurs and is linked to the outcome of infection by L. Viannia (asymptomatic, chronic or recurrent infection). This protocol is the first part of a series of studies that includes protocols 05-0139 and 06-0009. Specific objectives include: defining the expression of human inflammatory cytokines in the ex vivo recall response to live Leishmania for PBMCs of individuals presenting different clinical phenotypes at transcriptional, translational and secretion level; and assessing in situ and circulating cell populations from active, chronic and recurrent patients with respect to differentiation, activation, and co-activation markers. Patients (males and females) aged 18-70 years, with cutaneous leishmaniasis diagnosed in either Cali (CIDEIM) and/or Tumaco (San Andrés Hospital) on the Colombian Pacific Coast, and/or Chaparral, Tolima (San Juan Bautista Hospital) will be invited to participate in the study. Both historic (specific objective 1) and active (specific objective 2) patients will be enrolled. Asymptomatic individuals and healthy donors (controls) will also be invited to participate. Pregnant or breastfeeding women will not be enrolled. A total of 150 participants will be enrolled. For specific objective 1, participants will be asked to provide relevant demographic, clinical and epidemiologic information that will be recorded in a form designed for this purpose. They will also provide blood samples that will be analyzed to determine and compare the expression of human inflammatory cytokines in the ex vivo recall response to live Leishmania of PBMCs between the four groups. Specific objective 2 will be developed in CIDEIM-Cali, only. Participants will be asked to provide skin biopsies in addition to blood samples and relevant information. They will also undergo a skin blister procedure. Samples will be analyzed to characterize and compare in situ and circulating cell populations between the groups. Up to three visits are planned for this objective. The first visit will have a duration of up to 5 hours and the second one will have a duration of 30 minutes. A third visit may be programmed 48h-72h after the second visit for participants undergoing biopsy/skin blister procedure in order to evaluate possible bacterial superinfection and prevent complications. This visit will have a duration of 20 minutes. All visits will take place in a period of 4-5 days. In order to define the expression of human inflammatory cytokines in the ex vivo recall response to live Leishmania for PBMCs of individuals presenting different clinical phenotypes at transcriptional, translational and secretion level, the following variables will be measured and compared among the different groups: levels of expression of transcription factors in cells that have and have not been stimulated by live Leishmania; cytokine concentration at the transcriptional, and secretion levels in cells that have and have not been stimulated by live Leishmania; and percentage of specific PBMCs producing intracellular cytokines at translational level. In order to assess in situ (biopsy and blister) and circulating cell populations from active, chronic and recurrent patients with respect to differentiation, activation, and co-activation markers, the following variables will be measured and compared among the different groups: percentage of infiltrating leukocytes in blister fluid and biopsy, and circulating leukocytes in blood, expressing specific differentiation, activation and co-stimulation markers; mean fluorescence intensities of cells in blood, blister fluid, and biopsy expressing specific differentiation, activation and co-stimulation markers; percentage of specific cells from blister fluid, biopsies and blood producing intracellular cytokines IFN-gamma, IL-10, IL-4 and IL-13; and cytokine concentration in blister fluid.

ELIGIBILITY:
Inclusion Criteria:

All Groups:

- Age between 18-70 years

Inclusion Criteria for the 4 groups for specific objective 1:

Historical cases of chronic disease:

* Historic parasitologically confirmed, skin test positive CL patients who presented chronic CL lesions of > 6 months duration at the time of diagnosis.
* No active lesions
* Voluntary participation in the study
* Informed consent for HIV testing and participation in the study

Historical cases of recurrent disease:

* Historic CL patients who have developed new parasitologically confirmed lesions after resolution of prior disease
* No active lesions
* Voluntary participation in the study
* Informed consent for HIV testing and participation in the study

Asymptomatic infection cases:

* Resident of endemic area
* PBMCs responsive to leishmanial antigen in culture
* No history or evidence of active or prior dermal leishmaniasis
* Voluntary participation
* Informed consent for HIV testing and participation in the study

Healthy donors:

* No history or evidence of exposure to transmission of leishmaniasis
* Voluntary participation
* Informed consent for HIV testing and participation in the study

Inclusion Criteria for the 2 groups for specific objective 2:

Chronic disease group:

* Parasitologically confirmed chronic CL lesions of > 6 months duration in skin test positive patients.
* Voluntary participation in the study
* Informed consent for HIV testing and participation in the study

Recurrent disease group:

* Patients who have developed new parasitologically proven lesions after resolution of prior disease
* Voluntary participation in the study
* Informed consent for HIV testing and participation in the study

Exclusion Criteria:

Exclusion criteria all groups:

* Immunosuppressive disease
* Pharmacotherapy with drugs that are immunosuppressive
* Allergy/sensitivity to lidocaine family anesthetics or to latex
* Pregnancy
* Breastfeeding
* Unwillingness to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Age between 18-70 years
    1. Historical and confirmed cases of chronic leishmaniais disease with no current leishmaniasis
    2. Historical cases of confirmed recurrent leishmaniasis disease 3 Asymptomatic infection cases: (Resident of endemic area, PBMCs responsive to leishmanial antigen)
    4. Healthy donors:
  * No history or evidence of exposure to transmission of leishmaniasis
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2006-12; Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Gore Saravia, Ph.D., Study Director — CIDEIM, Cali Colombia; Diane McMahon-Pratt, Ph.D., Principal Investigator — Yale University
Locations (1):
- Centro Internacional de Entrenamiento e Investigaciones Medicas, CIDEIM, Cali, Colombia